CLINICAL TRIAL: NCT02931890
Title: A Multicentre Randomised Phase II Trial of Neo-adjuvant Chemotherapy Followed by Surgery vs. Neo-adjuvant Chemotherapy and Subsequent Chemoradiotherapy Followed by Surgery vs. Neo-adjuvant Chemoradiotherapy Followed by Surgery in Resectable Gastric Cancer
Brief Title: Multicentric Randomised Trial for Resectable Gastric Cancer
Acronym: CRITICS-II
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M15CRI; NL 55436.031.015 (Registry Identifier: CCMO); 2015-004627-31 (EudraCT Number)
Record Dates: First submitted 2016-09-14; First posted 2016-10-13 (Estimated); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Gastric Cancer
Keywords: gastric cancer; radiotherapy; chemoradiotherapy
MeSH Terms: conditions — Stomach Neoplasms | interventions — Docetaxel; Oxaliplatin; Capecitabine; Gastrectomy; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- neo-adjuvant chemotherapy followed by surgery (Active Comparator): 4 courses of 3 weekly DOC followed by surgery
  Interventions: Drug: Docetaxel; Drug: Oxaliplatin; Drug: Capecitabine; Procedure: gastrectomy
- neo-adjuvant chemo and subsequent CRT followed by surgery (Active Comparator): 2 courses of 3 weekly DOC and subsequent CRT followed by surgery
  Interventions: Drug: Docetaxel; Drug: Oxaliplatin; Drug: Capecitabine; Procedure: gastrectomy; Radiation: radiotherapy of gastric cancer; Drug: Paclitaxel; Drug: Carboplatin
- neo-adjuvant chemoradiotherapy followed by surgery (Active Comparator): chemoradiotherapy followed by surgery
  Interventions: Procedure: gastrectomy; Radiation: radiotherapy of gastric cancer; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Docetaxel — 3 weekly course of docetaxel i.v in arm 1 and 2
  Other Names: Taxotere
  Arms: neo-adjuvant chemo and subsequent CRT followed by surgery; neo-adjuvant chemotherapy followed by surgery
Drug: Oxaliplatin — 3 weekly course oxaliplatin as a 2 hr i.v. in arm 1 and 2
  Other Names: Eloxatin
  Arms: neo-adjuvant chemo and subsequent CRT followed by surgery; neo-adjuvant chemotherapy followed by surgery
Drug: Capecitabine — oral capecitabine in arm 1 and 2
  Other Names: Xeloda
  Arms: neo-adjuvant chemo and subsequent CRT followed by surgery; neo-adjuvant chemotherapy followed by surgery
Procedure: gastrectomy — resection of gastric cancer after pre-operative chemotherapy for all arms
Radiation: radiotherapy of gastric cancer — 5 weeks of radiation, 5 times a week with a total of 45 Gy (in arm 2 and 3)
  Arms: neo-adjuvant chemo and subsequent CRT followed by surgery; neo-adjuvant chemoradiotherapy followed by surgery
Drug: Paclitaxel — 5 weeks of paclitaxel i.v once a week (in arm 2 and 3)
  Arms: neo-adjuvant chemo and subsequent CRT followed by surgery; neo-adjuvant chemoradiotherapy followed by surgery
Drug: Carboplatin — 5 weeks of carboplatin i.v once a week (in arm 2 and 3)
  Arms: neo-adjuvant chemo and subsequent CRT followed by surgery; neo-adjuvant chemoradiotherapy followed by surgery

SUMMARY:
The CRITICS-II trial aims to identify the optimal preoperative regimen in resectable gastric cancer by comparing three investigational treatment arms: chemotherapy vs. chemotherapy and subsequent chemoradiotherapy vs. chemoradiotherapy. The rationale behind this trial design is based on the following concepts:

* Preoperative treatment is associated with better patient compliance than postoperative regimens
* Preoperative treatment increases the likelihood of disease downsizing/downstaging and radical R0 resections
* Preoperative paclitaxel/carboplatin-based concurrent chemoradiotherapy and DOC chemotherapy are effective, feasible and safe regimens

ELIGIBILITY:
Inclusion Criteria:

* TNM 8th ed stage IB-IIIC gastric cancer (histologically proven); tumour bulk has to be in the stomach but may involve gastro-oesophageal junction
* WHO < 2
* Age ≥ 18 yrs
* Resectable adenocarcinoma of the stomach or gastro-oesophageal junction
* No prior abdominal radiotherapy
* Haematology: Hb ≥5.0 mmol/l; leukocytes≥3.0x109/l, neutrophils ≥1.5x109/l, thrombocytes ≥100x109/l
* Renal function: serum creatinine ≤1.25x ULN, creatinine clearance ≥ 50 ml/min (calculated by Cockcroft and Gault formula) Liver function: total bilirubin ≤1.5x ULN, alkaline phosphatase and ASAT/ALAT ≤ 3x ULN
* At staging laparoscopy (mandatory) obtained biopsies of suspected peritoneal lesions and/or substantial free peritoneal fluid if any should be pathologically proven tumor negative
* Written informed consent
* Expected adequacy of follow-up
* Caloric intake≥1500 kcal/day, verified by a dietician before registration.
* if caloric intake is < 1500 kcal/day or if bodyweight has decreased > 10% over the last 6 months or > 5% over the last month, dietary intervention such as oral nutritional support or enteral tube feeding is mandatory

Exclusion Criteria:

* T1N0 disease (assessed by endoscopic ultrasound)
* Distant metastases
* Inoperable patients; due to technical surgery-related factors or general condition
* Previous malignancy, except adequately treated non-melanoma skin cancer or in-situ cancer of the cervix uteri; in case of a previous other malignancy with a disease-free period≥5 years, inclusion can be accepted after consultation of the principal investigator
* Solitary functioning kidney that will be within the radiation field
* Major surgery within 4 weeks prior to study treatment start, or lack of complete recovery from the effects of major surgery
* Uncontrolled (bacterial) infections
* Significant concomitant diseases preventing the safe administration of study drugs or likely to interfere with study assessments
* Uncontrolled angina pectoris, cardiac failure or clinically significant arrhythmias
* Continuous use of immunosuppressive agents equivalent to >10 mg daily prednison
* Concurrent use of the antiviral agent sorivudine or chemically related analogues, such as brivudine
* Neurotoxicity > CTC grade 1
* Pregnancy or breast feeding
* Patients (M/F) with reproductive potential not implementing adequate contraceptive measures
* Gastric or gastro-esophageal stent within radiation field

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Estimated)
Dates: Start 2017-12-21 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Event-Free survival | 1 year
  Event-free survival will be measured by clinical outcome and CT-scan

SECONDARY OUTCOMES:
Time to Event (events: local recurrence, regional recurrence, local-regional recurrence or progression, distant recurrence, or death from any cause) | 1 year
  Interval between randomization and event measured by clinical outcome and CT scan
Time to recurrence (events: local recurrence, regional recurrence, local-regional recurrence or progression, distant recurrence) | 1 year
  Interval between randomization and recurrence determined by clinical outcome and CT scan
Toxicity | 1 year
  Number of patients with treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Marcel Verheij, MD, PhD, Principal Investigator — The Netherlands Cancer Institute
Locations (28):
- Netherlands (28):
  - Zuyderland Medisch Centrum, Sittard-Geleen, Limburg
  - Viecuri Medisch Centrum, Venlo, Limburg
  - Elkerliek, Deurne, North Brabant
  - Catharina Ziekenhuis, Eindhoven, North Brabant
  - Maxima Medisch Centrum, Eindhoven, North Brabant
  - St. Anna Zorggroep, Geldrop, North Brabant
  - Elkerliek, Helmond, North Brabant
  - Instituut Verbeeten, Tilburg, North Brabant
  - Bernhoven, Uden, North Brabant
  - Maxima Medisch Centrum, Veldhoven, North Brabant
  - Spaarne Gasthuis, Hoofddorp, North Holland
  - Ziekenhuisgroep Twente, Almelo, Overijssel
  - Deventer Ziekenhuis, Deventer, Overijssel
  - Medisch Spectrum Twente, Enschede, Overijssel
  - Medisch Centrum Leeuwarden, Leeuwarden, Provincie Friesland
  - Radiotherapeutisch Instituut Friesland, Leeuwarden, Provincie Friesland
  - Reinier de Graaf Gasthuis, Delft, South Holland
  - Leids Universitair Medisch Centrum, Leiden, South Holland
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Netherlands Cancer Instituut, Amsterdam
  - Academisch Medisch Centrum, Amsterdam
  - Rijnstate, Arnhem
  - Ziekenhuis Gelderse Vallei, Ede
  - Universitair Medisch Centrum Groningen, Groningen
  - Ziekenhuis St Antonius, Nieuwegein
  - HAGA ziekenhuis, The Hague
  - Elisabeth Tweesteden Ziekenhuis, Tilburg
  - Universitair Medisch Centrum Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Slagter AE, Jansen EPM, van Laarhoven HWM, van Sandick JW, van Grieken NCT, Sikorska K, Cats A, Muller-Timmermans P, Hulshof MCCM, Boot H, Los M, Beerepoot LV, Peters FPJ, Hospers GAP, van Etten B, Hartgrink HH, van Berge Henegouwen MI, Nieuwenhuijzen GAP, van Hillegersberg R, van der Peet DL, Grabsch HI, Verheij M. CRITICS-II: a multicentre randomised phase II trial of neo-adjuvant chemotherapy followed by surgery versus neo-adjuvant chemotherapy and subsequent chemoradiotherapy followed by surgery versus neo-adjuvant chemoradiotherapy followed by surgery in resectable gastric cancer. BMC Cancer. 2018 Sep 10;18(1):877. doi: 10.1186/s12885-018-4770-2. PMID 30200910